CLINICAL TRIAL: NCT03314870
Title: Development of a Response Signature to Neoadjuvant Chemotherapy for Breast
Brief Title: Development of a Response Signature to Neoadjuvant Chemotherapy for Breast Cancer
Acronym: Breast-sign
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/25JUL/376
Record Dates: First submitted 2017-09-23; First posted 2017-10-19 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrospective study (Other): Tumoral tissue of 100 patients with breast cancer treated with neoadjuvant chemotherapy.
  Interventions: Genetic: Genetic signature
- Prospective study (Other): Tumoral tissue and plasma of 120 patients with breast cancer treated with neoadjuvant chemotherapy.
  Interventions: Genetic: Genetic signature

INTERVENTIONS:
Genetic: Genetic signature — To identify molecular signatures of EMT / immune status by using the random forest algorithm. The best signature will be measured by RT-qPCR and/or CATS-RNASeq technics.

SUMMARY:
Breast cancer is the most frequent cancer in women. It is often treated with neoadjuvant chemotherapy, administered before surgical resection. Unfortunately, many patients do not respond to this treatment, or only respond partially. Clinicians therefore need predictive biomarkers of treatment response. Thanks to an innovative technique, called CATS, this study aims at identifying blood and tissue biomarkers which are predictive of response to chemotherapy.

DETAILED DESCRIPTION:
Breast cancer is the most frequent cancer in women. It is often treated with neoadjuvant chemotherapy, administered before surgical resection. Unfortunately, many patients do not respond to this treatment, or only respond partially. Clinicians therefore need predictive biomarkers of treatment response. Thanks to an innovative technique, called CATS, this study aims at identifying blood and tissue biomarkers which are predictive of response to chemotherapy.

The objective of this study is to develop molecular signatures predictive of response to neoadjuvant chemotherapy which would be able to discriminate between patient groups based on their epithelio-mesenchymal transition (EMT) status and their immune status. As these two parameters are known to be responsible for incomplete responses to chemotherapy, investigators hypothesize that these signatures will be predictive of response to neoadjuvant chemotherapy. In a second step, researchers will evaluate the ability of these signatures to predict treatment response in breast cancer patients treated with neoadjuvant chemotherapy.

The investigators will investigate two types of signatures: a tissue signature and a circulating signature. The former is based on the level of expression of several mRNA and miRNA assessed by CATS-RNASeq in the biopsy. The circulating signature will be based on the expression level of several miRNA by the same technique. Given that the expression level of tumoral miRNA is affected by the EMT and immunological status, and given that tumors secrete miRNA in the circulation, investigators expect the miRNA plasma content to reflect the EMT and immunological status of the tumor. The circulating signature will have the additional advantage of being independent of tumor heterogeneity.

ELIGIBILITY:
Inclusion Criteria:

* Women and men with breast cancer
* Treated with neoadjuvant chemotherapy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of molecular signatures predictive of response to neoadjuvant chemotherapy which would be able to discriminate between patient groups based on their epithelio-mesenchymal transition status and their immune status. | an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: François DUHOUX, MD, PhD, Principal Investigator — francois.duhoux@uclouvain.be
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
There is no IPD